CLINICAL TRIAL: NCT03122847
Title: The Effect of 4.5 Gram Methylprednisolone Administered Once Weekly for 12 Weeks on Bone Metabolism in Graves´ Ophthalmopathy
Brief Title: Glucocorticoids and Bone in Graves' Ophthalmopathy
Status: Completed | Type: Observational
Sponsor: Torben Harsløf (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Torben Harsløf, MD, PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: GRO-BONE1
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples stored at -80C for batch analysis at study completion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: 30 patients with Graves' ophthalmopathy in which treatment with intravenous methylprednisolone is indicated
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Intravenous methylprednisolone
  Other Names: Solu Medrol

SUMMARY:
Continuous use of systemic glucocorticoids decreases bone mineral density and increases fracture risk. Graves' orbitopathy is treated with weekly infusion of high-dose intravenous glucocorticoid. The investigators aim at investigating whether this treatment regimen also affects bone metabolism.

DETAILED DESCRIPTION:
Systemic glucocorticoid increases bone resorption and decreases bone formation and thereby decreases bone mineral density and increases fracture risk. This effect is evident with a daily dose of 5 mg for three months or an accumulated dose of 450mg. There is, however, less evidence that intermittent use of glucocorticoids is harmful to bone.

Graves orbitopathy is treated with a weekly infusion of the glucocorticoid methylprednisolone and the accumulated dose over a 12-week course sums up to 4,500mg.

The investigators therefore want to investigate if that treatment regimen affects bone turnover, bone mineral density, or bone structure in 30 patients with Graves' orbitopathy.

ELIGIBILITY:
Inclusion Criteria:

* Graves Ophthalmopathy that requires treatment with intra-venous methylprednisolone

Exclusion Criteria:

* Treatment with osteoporosis medication
* Primary hyperparathyroidism
* Hypoparathyroidism
* Vitamin D < 20mmol/L
* Estimated glomerular filtration rate < 30 mL/min
* Liver disease
* Peroral treatment with glucocorticoids within last three months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 adult patients with Graves' Ophthalopathy
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torben Harsløf, MD, PhD, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus C, Central Jutland
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients: 32 patients with Graves' ophthalmopathy in which treatment with intravenous methylprednisolone is indicated
  Methylprednisolone: Intravenous methylprednisolone
Period: Overall Study
Arm/Group | Patients
Started | 39
Completed | 32
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Patients
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 32
Lumbar spine bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 1.0 (0.15)
Femoral neck bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 0.78 (0.11)
Total hip bone mineral density [Mean (Standard Deviation); unit: g/cm2] | 0.91 (0.13)
Tri-iodothyronine [Mean (Standard Deviation); unit: nmol/L] | 1.92 (0.67)
Thyroxine [Mean (Standard Deviation); unit: nmol/L] | 90.4 (35.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change Lumbar Spine Bone Mineral Density
Description: Percent change in lumbar spine bone mineral density from baseline to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Patients
Number analyzed (Participants) | 32
Percentage change | 1.37 (4.52)

2. Secondary Outcome: Percent Change Femoral Neck Bone Mineral Density
Description: Percent change in femoral neck bone mineral density from baseline to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Patients
Number analyzed (Participants) | 32
Percentage change | -0.32 (4.75)

3. Secondary Outcome: Percent Change Total Hip Bone Mineral Density
Description: Percent change in total hip bone mineral density from baseline to week 12
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Patients
Number analyzed (Participants) | 32
Percentage change | -0.18 (2.62)

4. Secondary Outcome: Bone Resorption
Description: Change in bone resorption measured by the biochemical marker C-terminal telopeptide of type 1 collagen (CTx) where higher measures show increased bone resorption that decreases bone mineral density and strength.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Patients
Number analyzed (Participants) | 32
microgram/L | -0.27 (0.32)

5. Secondary Outcome: Bone Formation
Description: Change in Bone Formation Measured by the Biochemical Marker procollagen type I N-propeptide (P1NP) where higher measures in combination with increased CTx (see measure 4) show increased bone resorption that decrease bone mineral density and strength but where lower levels may suggest decreased bone formation that may alsodecrease bone mineral density and strength.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: microgram/L
Arm/Group | Patients
Number analyzed (Participants) | 32
microgram/L | -52.3 (97.5)

6. Secondary Outcome: Percent Change in Bone Structure at the Radius
Description: Percent change in radial cortical volumteric BMD measured by high-resolution peripheral quantitative computed tomography
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Patients
Number analyzed (Participants) | 32
Percentage change | 0.98 (0.38)

7. Secondary Outcome: Percent Change in Bone Structure at the Tibia
Description: Percent change in tibial cortical volumetric BMD measured by high-resolution peripheral quantitative computed tomography
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Patients
Number analyzed (Participants) | 32
Percentage change | 1.35 (0.5)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Patients
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
Follow up corresponds to the treatment length of the disease but may have been too short to fully elucidate the effect of treatment on bone mass and structure. Moreover, the study design does not allow distinction of the effect of treatment with methylprednisolone and treatment of the underlying disease on bone.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03122847/Prot_SAP_000.pdf